CLINICAL TRIAL: NCT03294304
Title: BLASST-1 (Bladder Cancer Signal Seeking Trial): Phase II Trial of Neoadjuvant Nivolumab With Cisplatin and Gemcitabine in Muscle-Invasive Bladder Cancer (MIBC) Patients Undergoing Radical Cystectomy
Brief Title: BLASST-1 (Bladder Cancer Signal Seeking Trial): Nivolumab, Gemcitabine, and Cisplatin in Treatment of Muscle Invasive Bladder Cancer (MIBC) Undergoing Cystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017LS039
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: MIBC; UC; Immunotherapy; Bladder Cancer; Neoadjuvant; Nivolumab; Cisplatin; Gemcitabine
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab, Cisplatin, & Gemcitabine (Experimental)
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be given at a fixed dose of 360 mg IV over 30 minutes on Day 8 every 21 days for 4 cycles.
  Other Names: Opdivo
Drug: Cisplatin — Cisplatin will be given at 70 mg/m2 IV over 30 minutes on Day 1 every 21 days, and based on treating physician's discretion, split-dose cisplatin can be given at 35 mg/m2 IV Day 1 and Day 8 every 21 days for 4 cycles.
  Other Names: Platinol
Drug: Gemcitabine — Gemcitabine will be given at 1000 mg/m2 IV over 30 minutes on days 1, 8, and every 21 days for 4 cycles.
  Other Names: Gemzar

SUMMARY:
This is a multi-center Phase II study to determine the safety and efficacy of nivolumab when given in combination with cisplatin and gemcitabine as neoadjuvant treatment in patients with muscle-invasive bladder cancer (MIBC) prior to standard of care radical cystectomy. Patients will receive neoadjuvant treatment with nivolumab in combination with gemcitabine-cisplatin (GC) every 3 weeks for 4 treatment cycles over 12 weeks followed by standard of care radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MIBC (predominantly urothelial carcinoma) with clinical stage T2-T4a and N<1 disease (solitary lymph node measuring < 2 cm) and M0 and deemed eligible for radical cystectomy.
* Age ≥ 18 years
* ECOG Performance Status of 0 or 1.
* Required initial laboratory values within 14 days of study enrollment:

  * Absolute Neutrophil Count ≥ 1500 cells/mm^3
  * Platelets ≥ 100,000 cells/mm^3
  * Hemoglobin ≥ 9.0 g/dL
  * Bilirubin ≤ 1.5 times the upper limit of normal (ULN) for the institution (For patients with known Gilbert's disease: bilirubin ≤ 3 x ULN)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN for the institution
  * Creatinine clearance ≥ 50 ml/min by Cockcroft-Gault formula or 24 hour urinary clearance (CrCl = [140-age (years)] x actual weight (kg) / [72 x serum Cr (mg/dL)] (if patient is female multiply the above by 0.85) or 24 hour urinary creatinine clearance.
  * Alkaline phosphatase ≤ 2.5 x ULN for the institution
  * INR and aPTT ≤ 1.5 x ULN if not on therapeutic anticoagulation. Patients receiving therapeutic anticoagulation will be allowed if maintained on a stable dose.
* Females of childbearing potential and males who are not surgically sterile and with partners of childbearing potential must agree to use effective contraception during study treatment for 5 months for females and 7 months for males after the last dose of nivolumab.
* Ability to provide a signed and dated consent or have a legally authorized representative to provide written and signed consent prior to the initiation of any research related procedures.
* Patient must agree to submission of archived tumor (20-25 formalin-fixed paraffin embedded (FFPE) slides of 5-10 microns in thickness) from TURBT and radical cystectomy tissues. If archived samples are not available fresh tissue will be used.
* Ability to provide written consent prior to the initiation of any research related procedures.

Exclusion Criteria:

* Presence of N2-3 or M1 disease.
* Ineligible to receive cisplatin by meeting one or more of the following criteria;

  * Creatinine clearance of < 50 mL/min
  * Hearing loss of 25 dB at two contiguous frequencies with testing required if a patient has hearing loss - At the investigator's discretion, and after discussion with the patient, this exclusion may be waived if the potential benefit of cisplatin therapy is felt to outweigh the risk of further hearing loss.
  * CTCAE v4 Grade 2 or higher peripheral neuropathy,
  * New York Heart Association Class III or IV heart failure
  * ECOG performance status 2 or higher.
* Prior systemic therapy (intravenous) is not permitted. Prior intravesical therapies including intravesical gemcitabine is permitted for non-muscle invasive disease (i.e. T1 or lower).
* Prior treatment with cisplatin for bladder cancer.
* Prior treatment with anti-PD-1, CTLA-4, or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
* Prior therapeutic radiation to the bladder.
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure (>New York Heart Association Class 2), stroke, serious cardiac arrhythmia.
* Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness.
* Pregnancy, lactation, or breast-feeding. Women of childbearing potential must have a negative urine pregnancy test at screening.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, vascular thrombosis associated with antiphospholipid syndrome, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, systemic vasculitis, or glomerulonephritis.
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan, history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active hepatitis B virus (HBV, chronic or acute, defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C antibody. Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to Cycle 1, Day 1 and confirmed to be negative. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Active tuberculosis or BCG infection
* Active infection requiring systemic antibiotics for more than 7 days within 3 days prior to Cycle 1, Day 1. Prophylactic short-term antibiotics will be allowed.
* Administration of intravesical bacillus Calmette-Guerin (BCG) within 4 weeks before Cycle 1, Day 1
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study.
* Persisting toxicity from prior therapy (NCI CTCAE v4.03 Grade >1); however alopecia or other Grade <2 AEs not constituting a safety risk, based on Investigator's judgement, are acceptable.
* History of or active bone marrow disorders expected to interfere with study therapy (e.g. acute leukemias, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma).
* Prior allogeneic stem cell or solid organ transplant.
* Known primary central nervous system (CNS) malignancy.
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted but patients with psoriasis require a baseline ophthalmologic exam to rule out ocular manifestations. Rash must cover less than 10% of body surface area (BSA) and must be well controlled at baseline and only requiring topical steroids.
* Any other chronic medical condition or psychiatric condition, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative therapy. Patients on androgen deprivation therapy as part of adjuvant therapy after radiation for prostate cancer or patients on adjuvant hormonal therapies for breast cancer will be allowed if they are being considered for curative intent for bladder cancer.
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]-a or interleukin [IL]-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
* Concomitant use of systemic corticosteroids at physiologic doses or <10 mg/day of prednisone or equivalent.
* Concomitant use of another investigational agent and/or treatment with an investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five halflives of the investigational product, whichever is longer).
* Use of bisphosphonate therapy for osteoporosis will be allowed if started prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Badrinath Konety, MD, MBA, Principal Investigator — Masonic Cancer Center, University of Minnesota; Shilpa Gupta, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota
  - Huntsman Cancer Institute - University of Utah Health, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 22
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 15
  Female | 26
  Unknown | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response Rate (PaR) at Time of Radical Cystectomy. PaR is Defined as Absence of Residual MIBC at Cystectomy in the Surgical Specimen (Pathologic Down-staging to ≤pT1pN0 Which Includes pT0, pT1, pTa and pTis)
Description: Incidence of Measurable Disease "pT" in the TNM staging system refers to the size and extend of the primary tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b. pTa refers to noninvasive papillary carcinoma. pTis refers to carcinoma in situ (CIS) or a "flat tumor" stage. pN refers to lymph nodes. N0 mans cancer has not spread to nearby lymph nodes.
Time Frame: Surgery Day 1
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 27

2. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin (Cycle 1)
Description: Count of participants with Adverse Events related to Nivolumab with Gemcitabine/Cisplatin
Time Frame: Treatment Day 1 of cycle 1
Population: 2 participants were not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 7

3. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin (Cycle 1)
Description: Count of participants with Adverse Events related to Nivolumab with Gemcitabine/Cisplatin
Time Frame: Treatment Day 8 of cycle 1
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 27

4. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin (Cycle 2)
Description: Count of participants with Adverse Events related to Nivolumab with Gemcitabine/Cisplatin
Time Frame: Treatment Day 1 of cycle 2
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 18

5. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin (Cycle 2)
Description: Count of participants with Adverse Events related to Nivolumab with Gemcitabine/Cisplatin
Time Frame: Treament day 8 of cycle 2
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 15

6. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin (Cycle 3)
Description: Count of participants with Adverse Events related to Nivolumab with Gemcitabine/Cisplatin
Time Frame: Treatment day 1 of cycle 3
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 16

7. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin (Cycle 3)
Description: Count of participants with Adverse Events related to Nivolumab with Gemcitabine/Cisplatin
Time Frame: Treatment day 8 of cycle 3
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 13

8. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin (Cycle 4)
Description: Count of participants with Adverse Events related to Nivolumab with Gemcitabine/Cisplatin
Time Frame: Treatment day 1 of cycle 4
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 8

9. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin (Cycle 4)
Description: Count of participants with Adverse Events related to Nivolumab with Gemcitabine/Cisplatin
Time Frame: Treatment day 8 of cycle 4
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 11

10. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin
Description: Incidence of Adverse Events
Time Frame: 30 Days +/- 7 Days after last chemotherapy
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 5

11. Secondary Outcome: Safety of Nivolumab With Gemcitabine/Cisplatin
Description: Incidence of Adverse Events
Time Frame: 4 weeks post radical cystectomy
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 24

12. Secondary Outcome: Count of Participants Experiencing Progression Free Survival (PFS)
Description: Count of participants experiencing Progression Free Survival (PFS)
Time Frame: Every 3 Months for 2 Years
Population: 2 participants are not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
Number analyzed (Participants) | 41
Participants | 36

ADVERSE EVENTS:
Time Frame: 120 days after last dose nivolumab
Arm/Group | Nivolumab, Cisplatin, & Gemcitabine
All-Cause Mortality (participants affected / at risk) | 7/43
Serious Adverse Events (participants affected / at risk) | 11/43
Other Adverse Events (participants affected / at risk) | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab, Cisplatin, & Gemcitabine (N=43)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab, Cisplatin, & Gemcitabine (N=43)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (12)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 12 (18)
Alkaline phosphatase increased (Investigations) | 6 (6)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 25 (61)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Anxiety (Psychiatric disorders) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 11 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Blurred vision (Eye disorders) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Cardiac troponin I increased (Investigations) | 1 (1)
Chills (General disorders) | 4 (4)
Cholesterol high (Investigations) | 3 (3)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 24 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Creatinine increased (Investigations) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 10 (12)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Edema limbs (General disorders) | 7 (8)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (1)
Fatigue (General disorders) | 30 (37)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (3)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 13 (29)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (11)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (4)
Hemoglobin increased (Investigations) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (20)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hypertension (Vascular disorders) | 15 (24)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (15)
Hypokalemia (Metabolism and nutrition disorders) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (22)
Hyponatremia (Metabolism and nutrition disorders) | 10 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7)
Hypothyroidism (Endocrine disorders) | 7 (9)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Infusion related reaction (General disorders) | 2 (3)
Infusion site extravasation (General disorders) | 2 (2)
Injection site reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Investigations - Other, specify (Investigations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 6 (8)
Memory impairment (Nervous system disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 31 (37)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 20 (40)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Papulopustular rash (Infections and infestations) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5)
Phlebitis (Vascular disorders) | 2 (2)
Platelet count decreased (Investigations) | 13 (19)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (13)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Superficial thrombophlebitis (Vascular disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (6)
Tinnitus (Ear and labyrinth disorders) | 10 (10)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 7 (7)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 9 (10)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 3 (4)
Uterine pain (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (10)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 5 (5)
White blood cell decreased (Investigations) | 18 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT03294304/Prot_SAP_000.pdf